CLINICAL TRIAL: NCT02821429
Title: Respiratory Weaning Following Cardiac Surgery. Potential Interest of Combined Thoracic Echography in the Characterization of the Failure Causes.
Brief Title: Respiratory Weaning Following Cardiac Surgery.
Acronym: ETCCCV
Status: Withdrawn | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/15/7850
Record Dates: First submitted 2016-06-28; First posted 2016-07-01 (Estimated); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Respiratory Insufficiency
Keywords: Respiratory weaning; Pulmonary ventilation
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient with mechanical ventilation: Patient will be followed with combined Thoracic Echography Record
  Interventions: Other: Combined Thoracic Echography Record

INTERVENTIONS:
Other: Combined Thoracic Echography Record — This examination will be done to do the longitudinal follow-up of the patient

SUMMARY:
Respiratory weaning failure worsens prognostic of patients following on-pump cardiac surgery. There are increasing evidences that pulmonary, diaphragmatic or cardiologic echographies are useful in order to improve this critical medical status.

Based both on a previous study conducted in the critical care unit of Purpan and on literature we hypothesize that a combined thoracic echography score could be of interest. We make the hypothesis that the use of a score based on thoracic combined echography (ETC = cardiac, pulmonary and diaphragmatic) allows to predict the failure of respiratory weaning in cardiac surgery and allows to improve the characterization of the causes of this failure

ELIGIBILITY:
Inclusion Criteria:

* Adult (> 18 years old) beneficiating of mechanical ventilation following cardiac surgery
* Weaning test period
* Patient insured under the French social security system

Exclusion Criteria:

* Tracheostomy
* Neurological disorders
* Need for prophylactic non invasive ventilation.
* Global obstructive lung disease with a forced expiratory volume < 50%.
* Judicial protection
* Patient already included in a trial still running.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited during the pre anesthetic visit
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of predictive value of combined Thoracic Echography (ETC) as assessed by difference in the ETC score before and after extubation | 1 hour after the weaning test and 48h after

SECONDARY OUTCOMES:
Evaluation of predictive value of combined Thoracic Echography (ETC) as assessed T tube Test score difference between patient who succeed or failed the weaning test | H0 and 48h after the weaning test
Evaluation of diagnostic value of combined Thoracic Echography (ETC) after failure to weaning test as assessed be ECT scores collected | H0, H1 and H48

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas MAYEUR, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided